CLINICAL TRIAL: NCT06124612
Title: Assessing the Effect of Asundexian on Thrombotic Status, in Particular Endogenous Fibrinolysis, in Patients With Atrial Fibrillation
Brief Title: An Investigator-initiated Linked Study to OCEANIC-AF
Status: Recruiting | Type: Observational
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof Diana Gorog, Professor, University of Hertfordshire
Other Study IDs: RD2023-21
Record Dates: First submitted 2023-11-05; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Endogenous fibrinolysis; Global thrombosis test
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial fibrillation: Patients already enrolled in main OCEANIC-AF study.
  Interventions: Diagnostic Test: Thrombotic assessment

INTERVENTIONS:
Diagnostic Test: Thrombotic assessment — GTT
  The Global Thrombosis Test (GTT) (Thromboquest Limited, UK) is an in vitro method imitating high shear stress conditions akin to that which exist in a severely stenosed artery. The test measures platelet reactivity (occlusion time) and endogenous fibrinolysis time (lysis time).
  TEG Thromboelastography (TEG, Haemonetics Corporation, USA) is a technique that assesses the whole process of clotting and its viscoelastic properties, from the initial activation and aggregation of platelets, to the role of thrombin and finally the stability of the formed clot, as a measure of fibrinolytic resistance.
  Citrated plasma will be stored for subsequent evaluation of thrombosis and fibrinolysis markers (including but not restricted to D-dimer, PAI-1, hs-CRP, NETs)

SUMMARY:
Impaired endogenous fibrinolysis is a recently recognised risk factor for thrombotic events in patients with cardiovascular disease. Enhancing endogenous fibrinolysis in such individuals represents a way of reducing thrombosis risk. However, the optimal pharmacotherapy to enhance fibrinolysis is unclear.

The aim of this study is to assess the effect of asundexian on endogenous fibrinolysis and compare this to apixaban. If asundexian can enhance endogenous fibrinolysis, this could be used as targeted treatment for patients who despite optimal antithrombotic therapy, demonstrate impaired endogenous fibrinolysis.

DETAILED DESCRIPTION:
The risk of a clot forming in a blood vessel, which can cause a heart attack or stroke, is determined partly by how "sticky" the blood is and partly by the effectiveness of the natural defences in the blood in dissolving any clots that start forming (clot lysis, or "fibrinolysis"). There are available tests that can assess how "sticky" the blood is, and we can overcome that with specific blood-thinning medications (such as anticoagulants [such as warfarin, apixaban, rivaroxaban] and antiplatelet agents [such as aspirin and clopidogrel]). However, we have not been able to assess the effectiveness of natural clot dissolving mechanisms, until recently.

In the last few years, using new blood testing techniques, we and other groups, have shown that individuals who have less effective natural clot lysis, have a much higher risk of heart attack, stroke and death. Therefore, we would like to find medications that can make clot lysis more effective, in such individuals, to reduce their risk of stroke and heart attack. Unfortunately, most blood thinning tablets for long term use do not improve clot lysis.

Earlier, our group has shown that the anticoagulant apixaban, mildly improved clot lysis.

We would now like to assess clot lysis in patients taking apixaban and compare it to patients taking a very new type of anticoagulant called asundexian, to see if asundexian can improve clot lysis more than apixaban.

The easiest way to do this, is to test additional blood samples from patients who are already taking part in a clinical trial comparing apixaban and asundexian (OCEANIC-AF). OCEANIC-AF is a phase 3, multicentre, randomised clinical trial, comparing asundexian, a new type of blood thinner (factor XI inhibitor) with a commonly used blood thinner (apixaban, a factor X inhibitor), to see if it carries a lower risk of bleeding.

This is a prospective observational linked study to the main OCEANIC-AF study, to be undertaken in 2 centres in England. Patients enrolled in OCEANIC-AF at these 2 centres will have 4 additional blood samples taken, at baseline before starting the investigational drug or comparator, then at the 3, 6 and 12 month visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or over
2. Patients enrolled in OCEANIC-AF study
3. Free from the exclusion criteria below
4. The patient is willing and able to understand the Patient Information Sheet and provide written informed consent
5. The patient agrees to comply with the drawing of blood samples for the assessments.

Exclusion Criteria:

1. Inability to provide valid informed consent
2. Patients aged < 18 years of age
3. Patients with significant neurological, hepatic, renal, endocrine, gastrointestinal, pulmonary, haemorrhagic, metabolic or other disease likely to confound the study requirements or analyses
4. Patients with a history of substance abuse or signs or clinical features of active substance abuse or psychiatric disease
5. Alcohol consumption above 21 units per week
6. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study
7. Any major bleeding diathesis or blood dyscrasia (platelets <70 x 109/l, Hb <80 g/dl, INR >1.4, APTT >x 2 UNL, leucocyte count <3.5 x 109/l, neutrophil count <1 x 109/l)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients enrolled into OCEANIC-AF study at these two centres will be approached to also participate in this linked study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-03 (Estimated); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Thrombotic status | 12 months
  The main marker of interest is endogenous fibrinolysis time (LT)

CONTACTS AND LOCATIONS:
Overall Officials: Diana A Gorog, MD, PhD, Principal Investigator — East and North Hertfordshire NHS Trust
Locations (2):
- United Kingdom (2):
  - Liverpool Heart and Chest Hospital, Liverpool
  - East and North Herts NHS Trust, Stevenage